CLINICAL TRIAL: NCT04783948
Title: Validity and Reliability of the Turkish Version of the Pectus Carinatum Evaluation Questionnaire for Patients With Pectus Carinatum
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assistant Professor, Acibadem University
Other Study IDs: 2020-19/09
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Pectus Carinatum; Compliance; Brace
MeSH Terms: conditions — Pectus Carinatum; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Brace Treatment — Compliance to brace compression used for the correction of pectus carinatum will be evaluated.

SUMMARY:
Based on the hypothesis that the chest wall was still pliable in adolescence and could be reshaped in a normal position with the external suppressor applied on the chest, a pressure orthosis was started to be used in the pectus carinatum. It is the focus of attention as it is an alternative method to surgery for patients. However, the patient's compliance with the orthosis is difficult. Therefore, in our study, we aimed to investigate the Turkish Validity and Reliability of the Pectus Carinatum Evaluation Questionnaire, which is a questionnaire investigating the compliance with orthosis treatment in patients diagnosed with Pectus Carinatum by the doctor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with Pectus Carinatum by a doctor, have an orthosis indication (2 cm above the protrusion level) and who are given the orthosis for the first time
2. Having a correction pressure below 10 pounds per square inch (PSI) in the compression test
3. Between the ages of 10-18,
4. Having dissatisfaction with this defect

Exclusion Criteria:

1. Having severe scoliosis (Cobb angle over 20 degrees)
2. Having chronic systemic disease
3. Having a serious psychiatric illness
4. Having complex mixed type pectus deformity

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Pectus Carinatum
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Pectus Carinatum Evaluation Questionnaire | 15-21 days
  A questionnaire (Pectus Carinatum Evaluation Questionnaire, PCEQ) was developed by Pessanha et al to be applied in the follow-up of Pectus Carinatum patients. The PCEQ was divided into four different sections, allowing a thorough evaluation of compliance, symptoms, social influence and engagement with sports and daily activities.

SECONDARY OUTCOMES:
The Pectus Excavatum Evaluation Questionnaire | 15-21 days
  The Pectus Excavatum Evaluation Questionnaire (PEEQ) was developed and validated by Lawson et al to measure the physical and psychosocial quality-of-life changes after surgical repair of pectus excavatum. Each of the 17 items in the PEEQ is in a Likert scale format, where low scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Pectus Carinatum — https://www.nlm.nih.gov/